CLINICAL TRIAL: NCT01244087
Title: Pilot Clinical Trial (Phase II) of Inquiry-based Stress Reduction (IBSR) Program for Survivors of Breast Cancer
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Oncology Specialists, S.C. (Other)
Responsible Party: Sponsor
Other Study IDs: IBSR
Record Dates: First submitted 2010-11-09; First posted 2010-11-19 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Inquiry Based Stress Reduction
Keywords: Inquiry-based stress reduction; Quality of life; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The IBSR (Inquiry-based stress reduction) intervention, developed by Byron Katie (www.thework.com), trains subjects to reduce their perceived level of stress by self-inquiry of their thoughts and beliefs connected to stressful circumstances or symptoms. This meditative process, named "The Work", enables the participants to identify and question the stressful thoughts that cause their suffering. The core of IBSR is simply four questions and a turnaround, which is a way of experiencing the opposite of what the participant believes. This process is simple, powerful and can be easily implemented in daily life.

Therefore, on the basis of previous data and beneficial observations the investigators postulate that the clinical utility of IBSR mediation program may improve psychological and physical symptoms and quality of life among BC patients during the survivorship period. Thus, we will conduct a pilot/feasibility randomized controlled clinical trial designed to

* Assess feasibility of a IBSR intervention by examining attendance, drop-out rates, and program satisfaction.
* Determine whether IBSR intervention compared with usual care is efficacious in improving quality of life, psychological and physical status in BC survivors.

DETAILED DESCRIPTION:
Study methodology:

The proposed study is pilot/feasibility intervention study with pre and post measures. 30 participants will receive Inquiry-based stress reduction (IBSR) group intervention.

Population:

Women aged 21 or older previously diagnosed with Stage 0-III BC who underwent surgery and received adjuvant or neo-adjuvant chemotherapy and/or radiation will be recruited from the Tel Aviv Medical Center Oncology Department affiliated to Tel-Aviv university.

Inclusion Criteria:

1. Bx proven breast cancer
2. Known disease stage
3. Subjects completed treatment within the prior 18 months
4. Subjects are able to read and speak Hebrew at the ninth grade level or higher, as will be judged by their ability to complete a battery of self-report measures
5. Willing to sign an informed consent
6. Age 21-70

Exclusion criteria:

1. Stage IV BC,
2. Prophylactic mastectomy prior to the current treatment for BC,
3. Severe psychiatric diagnosis (e.g. bipolar disorder),
4. Treatment for recurrent BC

Data collection procedures:

1. Assessments will be taken at an initial baseline orientation and within 1 week at the end of the 12-week intervention
2. One week before IBSR classes will start, a baseline orientation will be held at this session, informed consent will be obtained, baseline data will be collected, and a brief overview of the IBSR program will be provided, which will highlight the 12-week class schedule
3. An additional assessment, will be collected 12 month after completion of group intervention

Intervention:

1. Subjects will receive weekly 3.5 hour sessions conducted by two facilitators trained in IBSR and certified by BKI to conduct this intervention.
2. Class size will range from 12-16 participants.
3. All the sessions will be standardized and follow the training manual developed to maintain consistency in the program.
4. Subjects will receive a training manual and CD's to support home practice of various forms of inquiry practices.
5. The training manual will include weekly exercises, and program content related to the content identified below. In addition, the manual will include a weekly diary for recording homework practice activities.

The IBSR-BC program is a 12-week program adapted for consideration of BC survivors' health status. During the process, participants will be encouraged to identify and inquire about their stressful thoughts: regarding relationships with others, Beliefs that prevent them to promote their health, Judgments regarding their body, cancer related stressful thoughts, self judgments, and fear from cancer recurrence, death and suffering. This intervention provides for management of specific emotional/psychological symptoms (stress, anxiety, depression, fatigue, and fear of recurrence) and physical symptoms, such as pain and sleep and enables the participants to inquire and be relieved of their stressful thoughts, and emotions caused by these thoughts. Through the use of self-inquiry practices subjects are taught to increase awareness of their thoughts and feelings, to observe their emotional and physical responses during situations perceived by them as stressful, and allow their mind to return to its true, peaceful, creative nature. Through the process of self inquiry, subjects take an active role in investigating their stressful thoughts, and by this regulating their stress and managing symptoms and emotions, thus enabling them to cope better with the distress of having cancer.

Throughout the 12-week IBSR(BC) program, all subjects will be requested to formally meditate and perform self inquiry exercises alone or with a partner for a minimum of 15-45 min per day, 6 days per week; this time increases per week as participants becomes more experienced.

Daily practice will be recorded in a diary and IBSR worksheets each day. Indicators of IBSR (BC) 'compliance' will be established at prior to 70% attendance at the IBSR(BC) sessions and completion of 70% of the homework assigned based on a minimum of 15-45 min practiced each day. The total number of minutes/hours practiced over the 6-week program will also be assessed.

Instruments and outcome measures:

Measures of health status before and at the end of the study (12 weeks) will include psychological status and quality of life subscales of physical and emotional health:

1. Health-related quality of life will be measured by the Functional Assessment of Cancer Therapy-Breast scale (FACT-B); it consists of the following subscales: physical well-being (PWB), social/family well-being (SWB), emotional well-being (EWB), functional well-being (FWB), and a breast cancer subscale (BCS). Overall scores range from 0-144 where a higher score indicates better health-related quality of life .
2. Perceived stress will be measured by the 10-item Perceived Stress Scale, which assesses how often in the past month one appraises life situations as being stressful; higher scores indicate more stress .
3. Level of fatigue will be measured by FACT-Fatigue, a 13-item validated instrument developed for assessment of fatigue in people with cancer. Responses are made on a 5-point Likert scale .
4. Depression will be evaluated by the Center for Epidemiologic studies-depression scale (CES-D). The CES-D is a 20-item self-report measure developed to screen for depressive symptoms. Scores range from 0 to 60, with higher scores indicating more symptoms of depression .
5. Spiritual well-being will be assessed by FACIT-Spirituality (FACIT-Sp), a 12-item spirituality scale assesses. This scale has two domains, sense of meaning/peace (8 items) and role of faith (4 items). Higher scores indicate higher levels of spirituality .
6. Sleep quality will be measured by the Pittsburgh sleep quality inventory (PSQI). The PSQI is a reliable 19-item self-report measure to assess subjective sleep quality in the past month. It measures: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction .

Clinical data will be obtained from chart reviews conducted by a research nurse. Standard demographic data will be collected along with a detailed clinical history form completed by self-report and chart review to document prior medical history, lifestyle behaviors (e.g. smoking and exercise), and concomitant medication use. For this analysis, all measures of physical and psychological status will be treated as co-equal outcomes.

Statistical methods The intent to treat principle will be used for all analyses. Baseline data will be compared between the two groups by use of chi-square tests for categorical variables and Student t test for continuous variables. Analysis of covariance (ANCOVA) mixed models will be used to examine differences in post intervention scores from baseline, adjusting for baseline value of each outcome variable. All outcome measures will be analyzed separately, with a p-value p <0.05 indicating statistical significance (measures with p-values 0.05<p< 0.10 will be noted, as a trend towards significance may exist).

ELIGIBILITY:
Inclusion Criteria:

1. Bx proven breast cancer
2. Known disease stage
3. Subjects completed treatment within the prior 18 months
4. Subjects are able to read and speak Hebrew at the ninth grade level or higher, as will be judged by their ability to complete a battery of self-report measures
5. Willing to sign an informed consent
6. Age 21-70

Exclusion Criteria:

1. Stage IV BC
2. Prophylactic mastectomy prior to the current treatment for BC
3. Severe psychiatric diagnosis (e.g. bipolar disorder)
4. Treatment for recurrent BC

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 21 or older previously diagnosed with Stage 0-III BC who underwent surgery and received adjuvant or neo-adjuvant chemotherapy and/or radiation will be recruited
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Ron, MD, Principal Investigator — Sourasky M.C.
Locations (1):
- Sourasky M.C.Oncology Department, Tel Aviv, Israel